CLINICAL TRIAL: NCT00174902
Title: The Effect of Beta-Blockers, Aspirin, and Natural Habituation on Procoagulant Activity, Expression of Cellular Adhesion Molecules, and Endothelial Activation in Response to Acute Mental Stress: a Randomized Controlled Trial.
Brief Title: The Effect of Beta-Blockers and Aspirin on Hemostasis and Endothelial Function After Acute Mental Stress
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Swiss National Science Foundation (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: SNF 32-68277
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2006-10-25 (Estimated); Status verified 2003-10

CONDITIONS: Arteriosclerosis; Stress, Psychological
Keywords: Randomized controlled trial; Blood platelets; Hemostasis; Stress, psychological; Adrenergic beta-antagonists; Aspirin; Endothelium; Arteriosclerosis
MeSH Terms: conditions — Arteriosclerosis; Stress, Psychological | interventions — Propranolol; Pharmaceutical Preparations; Aspirin

INTERVENTIONS:
Drug: inderal (drug), acetylsalicylic acid (drug)

SUMMARY:
This randomized double-blinded controlled trial uses a factorial design to investigate whether application of beta-blockers (inderal 80 mg) or aspirin (100 mg) or a combination thereof has an effect on the activation of the hemostatic system, the platelets and the endothelium in response to acute mental stress. Specifically we test the hypothesis that inderal attenuates the activation of the hemostatic system as compared to placebo. The second hypothesis is that aspirin attenuates the activation of platelets as compared to placebo. Subjects will be randomly allocated to either of the four following study arms: placebo - inderal - aspirin - inderal plus aspirin. Subjects will receive the study medication for five days prior to the mental stress. The acute mental stress consists of a public speaking session of 10 min duration immediately followed by a mental arithmetic test of 5 min duration. Blood will be collected prior to the stress, immediately thereafter, at 45 min at at 1 hour and 45 min.

DETAILED DESCRIPTION:
Background: Population based studies have established hemostatic abnormalities as independent risk factors for atherosclerosis and related adverse outcomes. These abnormalities are characterized as prothrombotic by elevated plasma levels of e.g. fibrinogen or D-dimer. Prothrombotic states appear to aggravate the impact of other risk factors, e.g. hypertension. Other epidemiologic studies have shown a sizable association between chronic mental stress (e. g. marital discord in women) or acute mental stress (anger) and coronary heart disease. A large case-crossover study attributed a 2.3-fold increased relative risk of acute myocardial infarction during the 2 hours following outbursts of anger. This risk was modified by aspirin (risk ratio of 2.9 in non-users, risk-ratio of 1.4 with prior to aspirin intake). We have recently shown that acute mental stress is followed by profound rises of D-dimer and induction of a prothrombotic state. In real life, individuals are frequently and repetitively exposed to similar stressors (e.g. work or marital discord). Those who fail to habituate and to mitigate their adrenergic responses and hemostatic changes, may be at increased risk of rapid progression of atherosclerosis. These individuals might particularly benefit from preventive medication with beta-blockers or aspirin.

Objectives: To elucidate whether administration of non-specific beta-blockers, aspirin or both may abrogate the prothrombotic shift in the hemostatic balance in response to acute mental stress.

To elucidate the pathway leading from central nervous system arousal after acute mental stress to increases in plasma D-dimer levels by investigating intermediate steps in the process, including activation of mononuclear and endothelial cells, of platelets, and of hemostatic factors.

To show that some individuals do not habituate when repetitively being exposed to the same stressor or/and that habituation blunts the stress response as do beta-blocking medication, aspirin or both.

Subjects: 80 healthy male and nonpregnant female non-smokers aged 40 - 55 years.

Methods: Randomized, double-blind, two-by-two factorial design. A public speaking stress will be applied in two different experiments. 1) The first experiment consists of a habituation study wherein 20 subjects will be stressed three times with intervals of 1 week apart. 2) The second experiment consists of a medication study wherein 60 individuals (other than those taking part in the habituation study) will be randomly assigned to one of the following four arms: 1) placebo/placebo, 2) placebo/beta-blocker, 3) placebo/aspirin, 4) beta-blocker/aspirin. Beta-blocker medication consists of 80 mg/day of propranolol (Inderal LA 80), aspirin will be given in a dose of 100 mg/day. Blood will be collected before, immediately after, and at 45 min, and at 1 hour and 45 min after the stress task in both experiments. In both experiments, subjects will be fully debriefed after the first stressor. The primary dependent variable is the change score of plasma levels of D-dimer after the stressor. Data will be analyzed by two-way ANOVA with the experimental condition being the first factor and with the experiment repetition being the second factor. Intermediate variables measured for elucidating the biological pathway leading to changes in D-dimer are: a) arousal of neuro-endocrine circuits: plasma levels of epinephrine and nor-epinephrine, salivary cortisol levels; b) activation / alteration of circulating mononuclear cells: quantitative determination of subpopulations by flow-cytometry, expression of L-selectin (CD62L), lymphocyte function associated antigen 1 (LFA-1), CD154 (expressed on activated T-lymphocytes), and tissue-factor on monocytes; c) activation of endothelial cells: plasma levels of soluble intercellular adhesion molecule 1 (sICAM-1), soluble vascular cellular adhesion molecule 1 (sVCAM-1), endothelin-1, and von Willebrand factor (vWF); d) balance between prothrombotic and fibrinolytic activity: plasma levels of D-dimer, fibrinogen, thrombin/antithrombin III complexes, tissue plasminogen activator, and plasminogen activator inhibitor-1.

ELIGIBILITY:
Inclusion Criteria:

* Life-time non-smoker or non-smoker for more than a year,
* native language Swiss-German,
* systolic blood pressure <160 mm Hg, diastolic blood pressure <100 mm Hg.
* Subjects must have a body mass index that is not considered to be a cardiovascular risk factor, i.e. ≤ 26.5 kg/m2.

Exclusion Criteria:

* Individuals reporting cardiovascular disease, renal disorders, endocrine disorders, hepatopathy, psychiatric disorders or who take regular medication for any of these conditions.
* Persons are excluded, who report to drink >5 cups (0.15 l each) of brewed coffee (> 500 mg caffeine) a day, or who report drink more than 1.0 l beer and 0.45 l wine per day, respectively.
* All subjects on regular beta-blocking or aspirin medication are excluded from the study.
* Participants will be required not to take aspirin or any other non-steroidal anti-inflammatory drug during the study period, beginning 10 days prior to the first study medication.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80
Dates: Start 2003-10; Study Completion 2004-08

PRIMARY OUTCOMES:
Change scores in plasma levels of D-dimer determined by subtracting levels immediately after the stressor as compared to baseline levels prior to the stressor.

SECONDARY OUTCOMES:
Change scores of a) monocyte and T-lymphocyte expression of L-selectin, lymphocyte-function associated antigen (LFA-1), and CD40L
monocyte tissue-factor antigen (CD 142) expression
plasma levels of TAT, t-PA, and PAI-1
plasma levels of soluble intercellular adhesion molecule (sICAM-1), soluble vascular adhesion molecule (sVCAM-1), endothelin-1, and vWF

CONTACTS AND LOCATIONS:
Overall Officials: Joachim E Fischer, MD, MSc, Principal Investigator — Swiss Federal Institute of Technology, Institute of Behavioral Sciences
Locations (1):
- Institute of Behavioral Sciences, Swiss Federal Institute of Technology, Zurich, Switzerland

REFERENCES:
- [Background] von Kanel R, Mills PJ, Ziegler MG, Dimsdale JE. Effect of beta2-adrenergic receptor functioning and increased norepinephrine on the hypercoagulable state with mental stress. Am Heart J. 2002 Jul;144(1):68-72. doi: 10.1067/mhj.2002.123146. PMID 12094190
- [Result] Mischler K, Fischer JE, Zgraggen L, Kudielka BM, Preckel D, von Kanel R. The effect of repeated acute mental stress on habituation and recovery responses in hemoconcentration and blood cells in healthy men. Life Sci. 2005 Jul 22;77(10):1166-79. doi: 10.1016/j.lfs.2005.03.006. Epub 2005 Apr 26. PMID 15978266
- [Result] von Kanel R, Kudielka BM, Preckel D, Hanebuth D, Fischer JE. Delayed response and lack of habituation in plasma interleukin-6 to acute mental stress in men. Brain Behav Immun. 2006 Jan;20(1):40-8. doi: 10.1016/j.bbi.2005.03.013. PMID 15890495
- [Result] von Kanel R, Preckel D, Zgraggen L, Mischler K, Kudielka BM, Haeberli A, Fischer JE. The effect of natural habituation on coagulation responses to acute mental stress and recovery in men. Thromb Haemost. 2004 Dec;92(6):1327-35. doi: 10.1160/TH04-04-0223. PMID 15583741